CLINICAL TRIAL: NCT05496270
Title: Surgery Alone Versus Neoadjuvant Treatment Followed by Surgery For MRI-defined T3 Mid-low Rectal Cancer: A Retrospective Cohort Study
Brief Title: Surgery Alone Versus Neoadjuvant Treatment Followed by Surgery For MRI-defined T3 Mid-low Rectal Cancer
Status: Completed | Type: Observational
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Yanhong Deng, Professor, Sun Yat-sen University
Other Study IDs: GIHSYSU-28
Record Dates: First submitted 2022-08-09; First posted 2022-08-11 (Actual); Last update posted 2022-08-11 (Actual); Status verified 2022-08

CONDITIONS: Rectal Cancer
MeSH Terms: conditions — Rectal Neoplasms | interventions — Neoadjuvant Therapy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- TME: patients only underwent TME
  Interventions: Procedure: total mesorectal excision
- nCRT+TME: patients underwent TME following neoadjuvant treatment
  Interventions: Procedure: total mesorectal excision

INTERVENTIONS:
Procedure: total mesorectal excision
  Other Names: neoadjuvant treatment

SUMMARY:
Neoadjuvant treatments (nCRT) are becoming the standard treatment for patients with stage II or stage III mid-low rectal cancer. In fact, with the introduction of total mesorectal excision, the local recurrence has been reduced significantly. Recently few studies have shown that surgery alone is enough for patients with T3 rectal cancer. These issues raised the question of whether nCRT is needed for all T3 rectal cancer patients. Therefore, this study was designed to compare the long-term oncological outcomes between surgery and surgery following nCRT among patients with MRI-defined T3, clear MRF mid-low rectal cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Eighteen- to eighty-year-old patients.
2. T3 rectal cancer with clear mesorectal fascia (MRF),
3. within 12 cm from the anal verge at initial diagnosis by magnetic resonance imaging (MRI)

Exclusion Criteria:

1. emergency surgery due to bleeding, perforation, and bowel obstruction,
2. recurrent rectal cancer,
3. inflammatory bowel disease,
4. Stage IV.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: T3 mid-low rectal cancer patients with clear MRF
Sampling Method: Non-Probability Sample
Enrollment: 1509 (Actual)
Dates: Start 2014-01 (Actual); Primary Completion 2019-01 (Actual); Study Completion 2022-08 (Actual)

PRIMARY OUTCOMES:
3-year diseases free survival | 3 years after surgery

SECONDARY OUTCOMES:
Margin-free （R0）resection rate | Immediately after the surgery
3-year overall survival rate | 3 years after surgery
Number of participants with surgical complications | 30 days after surgery
Local recurrence rate | 3 years after the surgery

IPD SHARING:
Plan to Share IPD: Undecided
The source data of the published results can be shared; they are available from the corresponding author upon reasonable request (kangl@mail.sysu.edu.cn).